CLINICAL TRIAL: NCT03857503
Title: Radiographic Imaging Validation and EvALuation for Angio iFR (ReVEAL iFR)
Acronym: ReVEAL
Status: Completed | Type: Observational
Sponsor: Volcano Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 180102
Record Dates: First submitted 2018-11-12; First posted 2019-02-28 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Cardiac Ischemia; Coronary Artery Disease; Coronary Stenosis
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary Lesion Assessment with iFR: Patients referred for cardiac catheterization for diagnostic and/or treatment purposes will undergo a screening angiogram to assess eligibility. Eligible patients will be those with at least one major epicardial vessel having a lesion of 40-90% diameter stenosis per visual assessment of angiogram.
  Interventions: Diagnostic Test: iFR

INTERVENTIONS:
Diagnostic Test: iFR — Patients will undergo standard of care diagnostic coronary angiography using established invasive physiological criteria for iFR and FFR to aid in clinical decision making for coronary revascularization.
  Angiograms will be made in at least two projections, and the treating physician will record his/her estimation of stenosis severity.
  Resting iFR and Pd/Pa measures will then be made distal to the target lesion; adenosine will be administered, and the FFR measures will be made without moving the wire. An iFR pullback will then be made after hyperemia as abated. Patients will be treated or deferred from treatment based on physician decision aided by the iFR measures.

SUMMARY:
The Philips Angio-iFR medical software device is intended to provide information on the functional significance of a coronary artery lesion to provide guidance on diagnostic decisions similar to that obtained through invasive measures of iFR and FFR. The software application uses the vessel geometry obtained from a coronary angiographic image together with a lumped parameter physiological model to provide the associated iFR and FFR estimates.

DETAILED DESCRIPTION:
This study is intended to demonstrate the diagnostic performance of the image-derived physiology model using the invasive physiological measures as the reference standard.

Specific objectives include the following:

i) Demonstrate the sensitivity and specificity of image-derived iFR and FFR results for identifying functionally significant lesions as determined by the corresponding invasive measures; ii) Demonstrate the diagnostic agreement of image-derived iFR and FFR estimates with the corresponding invasive measures; iii) Demonstrate the diagnostic performance of image derived physiology estimate (iFR/FFR) is superior to visual angiographic assessment for the identification of functionally significant stenoses as determined by the corresponding invasive physiology measures; iv) Demonstrate reproducibility of the image-derived estimate for a given operator and across multiple operators for a given lesion.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old
2. At least 1 de-novo lesion in 1 or more major epicardial vessels of 40-90% angiographic stenosis with a reference vessel size ≥2.5mm in the diseased segment by visual estimate
3. Able and willing to provide informed consent

Exclusion Criteria:

1. Presenting with an acute coronary syndrome (ACS), or documented ACS within 4 weeks prior to the scheduled index procedure
2. Cardiogenic shock (sustained (>10 min) systolic blood pressure <90 mmHg in absence of inotropic support or the presence of an intra-aortic balloon pump)
3. Presence of cardiac arrhythmias (e.g., atrial fibrillation, AV-block)
4. Prior cardiac surgery or implant, including CABG, heart transplant, surgical heart valve replacement or repair, TAVI/TAVR, presence of an ICD or pacemaker
5. Target vessel supplied by a left main coronary artery demonstrating any disease present (isolated or non-isolated)
6. Target vessel supplied by right coronary artery demonstrating any ostial disease (located immediately at the origin of the coronary vessels from the aorta)
7. Target vessel with Chronic Total Occlusion (CTO) in the ipsilateral territory or target vessel with an untreated CTO in the contralateral territory. Note: if a CTO existing in the contralateral territory is successfully opened, the target vessel in the contralateral territory can be included following CTO treatment.
8. Target vessel with severe tortuosity (≥1 bends of 90° or more, or ≥3 or more bends of 45°- 90° proximal to the diseased segment)
9. Target vessel with heavy calcification (multiple persisting opacifications of the coronary wall visible in more than one projection surrounding the complete lumen of the coronary artery at the site of the lesion.)
10. Target vessel with TIMI flow grade 1 or 0
11. Target vessel with severe diffuse disease (more than 75% of the length of the segment having a vessel diameter of 2mm, irrespective of the presence or absence of a lesion)
12. Target lesion is at a bifurcation/trifurcation
13. Target arteries supplying akinetic or severely hypokinetic territories if already known based on prior imaging
14. Target vessel is supplied by major collaterals
15. Target stenosis associated with myocardial bridge
16. Any vascular abnormality precluding optimal contrast opacification (e,g, thrombus, ulceration)
17. Severe aortic or mitral valve disease
18. Known ejection fraction ≤30%
19. Known severe renal insufficiency (eGFR<30ml/min/1.72m2)
20. Any fluoroscopic interference that renders the wire position unclear
21. Contraindication for adenosine or other hyperemic agent (e.g., caffeine ingestion ≤18 hours, COPD, hypotension, AV block)
22. Known pregnancy or planning to become pregnant
23. Participating in another interventional investigational study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for cardiac catheterization for diagnostic and/or treatment purposes will undergo a screening angiogram to assess eligibility. Eligible patients will be those with at least one major epicardial vessel having a lesion of 40-90% diameter stenosis per visual assessment of angiogram.
Sampling Method: Probability Sample
Enrollment: 441 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of the image-derived iFR | 1 day
  Diagnostic accuracy of the image-derived iFR and FFR estimate for a given lesion compared to the corresponding invasive iFR and FFR values.

CONTACTS AND LOCATIONS:
Locations (40):
- United States (19):
  - VA Medical Center, Long Beach, California
  - Colorado Heart and Vascular/St Anthony's, Lakewood, Colorado
  - Yale University Hospital, New Haven, Connecticut
  - Memorial Regional Hospital, Hollywood, Florida
  - Memorial Hospital- West, Pembroke Pines, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - Ascension St. John Hospital, Detroit, Michigan
  - Catholic Medical Center, Manchester, New Hampshire
  - South Side Hospital, Bay Shore, New York
  - University at Buffalo, Buffalo, New York
  - St Francis Hospital, Roslyn, New York
  - Duke University Hospital, Durham, North Carolina
  - NC Heart & Vascular, Goldsboro, North Carolina
  - Integris Heart Hospital, Oklahoma City, Oklahoma
  - Bryn Mawr Hospital, Wynnewood, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Centennial Heart, Nashville, Tennessee
  - Baylor Scott & White Research Institute, Dallas, Texas
- Germany (4):
  - Unversitatklinikum, Freiburg, Freiburg im Breisgau
  - Gemeinschaftsklinikum, Koblenz, Koblenz
  - Universitatklinikum, Mannheim, Mannheim
  - Robert-Bosch Krankenhaus, Stuttgart, Stuttgart
- University Hospital Galway, CRFG, Galway, Ireland
- Japan (3):
  - Gifu Heart Center, Gifu
  - Ehime Medical University, Matsuyama
  - Wakayama Medical University, Wakayama
- Netherlands (6):
  - AMC Amsterdam, Amsterdam
  - Amphia Ziekenhuis Breda, Breda
  - Medische Spectrum Twente, Enschede
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Sint Antonius Ziekenhuis, Nieuwegein
  - Radboud UMC, Nijmegen
- Spain (2):
  - Hospital Universitario de Léon, León
  - Hospital Clinico San Carlos, Madrid
- United Kingdom (5):
  - Basildon Univeristy Hospital, Basildon
  - Blackpool Victoria hospital, Blackpool
  - Royal Bournemouth hospital, Bournemouth
  - Imperial College of London- Hammersmith Hospital, London
  - University of Southampton, Southampton

REFERENCES:
- [Derived] Onuma Y, Ninomiya K, Sjauw K, Damman P, Matsuo H, von Birgelen C, Sevestre E, Ono M, O'Leary N, Garg S, van Lavieren MA, Inderbitzen B, Akasaka T, Escaned J, Patel MR, Serruys PW; ReVEAL iFR Investigators. Accuracy of instantaneous wave-free ratio and fractional flow reserve derived from single coronary angiographic projections. Am Heart J. 2025 Oct;288:111-121. doi: 10.1016/j.ahj.2025.03.001. Epub 2025 Mar 11. PMID 40081745
- [Derived] Revaiah PC, Tsai TY, Chinhenzva A, Miyashita K, Tobe A, Oshima A, Ferraz-Costa G, Garg S, Biscaglia S, Patel M, Collet C, Akasaka T, Escaned J, Onuma Y, Serruys PW. Physiological Disease Pattern as Assessed by Pull Back Pressure Gradient Index in Vessels With FFR/iFR Discordance. JACC Cardiovasc Interv. 2025 Apr 14;18(7):823-834. doi: 10.1016/j.jcin.2024.12.017. Epub 2025 Feb 19. PMID 39985510
- [Derived] Ono M, Serruys PW, Patel MR, Escaned J, Akasaka T, Lavieren MAV, Haase C, Grass M, Kogame N, Hara H, Kawashima H, Wykrzykowska JJ, Piek JJ, Garg S, O'Leary N, Inderbitzen B, Onuma Y. A prospective multicenter validation study for a novel angiography-derived physiological assessment software: Rationale and design of the radiographic imaging validation and evaluation for Angio-iFR (ReVEAL iFR) study. Am Heart J. 2021 Sep;239:19-26. doi: 10.1016/j.ahj.2021.05.004. Epub 2021 May 13. PMID 33992606